CLINICAL TRIAL: NCT03923348
Title: Pelvic Floor Muscle Training With the Leva® System for Treatment of Urge Predominant Urinary Incontinence: A Pilot Study
Brief Title: Pelvic Floor Muscle Training With Leva System for Urge Incontinence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Recruitment and Re-prioritizing of Sponsor-funding
Sponsor: The Christ Hospital (Other)
Collaborators: Renovia, Inc. (Industry)
Responsible Party: Principal Investigator, Anne Stachowicz, Fellow Physician, The Christ Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-71
Record Dates: First submitted 2019-03-18; First posted 2019-04-22 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Overactive Bladder; Urge Urinary Incontinence; Mixed Urinary Incontinence
Keywords: female urinary incontinence; urge urinary incontinence; urgency; frequency; overactive bladder; pelvic floor muscle training; biofeedback
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Intervention Model Description: Non-blinded non-comparative pilot trial in which subjects with pure urge urinary incontinence (UUI) or urge-predominant mixed urinary incontinence (U-MUI) who are candidates for pelvic floor physical therapy or other first line treatments for UUI/U-MUI use the leva® system twice-daily at home in addition to behavioral therapies for 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Leva Users (Experimental): Subjects with pure urge urinary incontinence (UUI) or urge-predominant mixed urinary incontinence (U-MUI) who are candidates for pelvic floor physical therapy or other first line treatments for UUI/U-MUI use the leva® system twice-daily at home in addition to behavioral therapies for 8 weeks.
  Interventions: Device: Leva device

INTERVENTIONS:
Device: Leva device — The leva® Pelvic Digital Health System by Renovia Inc is a novel tool for subjects with urinary incontinence to train and strengthen pelvic floor muscles via directional mechano-transductive feedback on performance in the privacy of their own homes.

SUMMARY:
This is a pilot non-comparative study to assess the effectiveness of pelvic floor muscle training guided by the leva® system for improving change in subject-reported incontinence-related quality of life and urgency urinary incontinence (UUI) episode frequency based on voiding diaries in women at 8 weeks.

DETAILED DESCRIPTION:
Our study aims to investigate a new alternative to formal pelvic floor physical therapy that may provide subjects with a more accessible, private method of undergoing pelvic floor muscle training (PFMT) with real-time biofeedback on performance. The leva® Pelvic Digital Health System by Renovia Inc is a novel tool for subjects with urinary incontinence to train and strengthen pelvic floor muscles via directional mechano-transductive feedback on performance in the privacy of their own homes. We hypothesize that women using the leva® System will experience significant improvements in subjective urge-related incontinence symptoms. In addition, changes in incontinence-related quality of life and UUI episode frequency will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years old
* Urinary incontinence for ≥ 3 months
* Reporting at least "moderate bother" on Item 2 on the UDI-6, "Do you experience urine leakage in related to the feeling of urgency" (on new patient paperwork)
* If mixed urinary incontinence, Medical Epidemiologic Social Aspect of Aging Urinary Incontinence Questionnaire (MESA) score indicating urge-predominant MUI (Urge subscale % > Stress subscale %)
* Presence of ≥ 1 UUI episode on 3-d bladder diary (see Appendix 2)
* Is the baseline bladder diary consistent with the patient's typical habits?
* Not currently taking anti-muscarinic or beta3 agonist therapy (after at least 2 week wash-out period)
* Brink Score > 3 (see below)
* Access to smartphone technology, including iOS or Android™

Exclusion Criteria:

* Non-English speakers
* Severely impaired mobility or cognition
* Spinal cord injury or advanced/severe neurologic condition including Multiple Sclerosis, Parkinson's Disease
* Concomitant prolapse beyond the hymen or repair of prolapse in the previous 6 months
* Received intravesical botulinum injection within the previous 12 months
* History of implanted nerve stimulator for incontinence
* History of prior sling or vaginal mesh placement
* Previous diagnosis of Interstitial cystitis
* Active pelvic organ malignancy
* History of pelvic radiation
* Urethral obstruction
* Urinary retention or prolonged catheter use
* Less than 12 months post-partum are currently pregnant, or plan to become pregnant in the following 12 months
* Untreated symptomatic urinary tract infection
* Unevaluated hematuria
* Medical instability
* Not available for follow-up in 6 months
* Participation in other research trials that could influence results of this study

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-06-06 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
Urogenital Distress Inventory | Change from Baseline UDI score to 8 weeks and 6 months post-intervention
  The Urogenital Distress Inventory (UDI) is a 19-item questionnaire assessing subjective symptoms of pelvic floor disorders including incontinence. The 19 items fall into one of three subscales (Irritative symptoms, Obstructive symptoms, and Stress Symptoms). . The subject responds to each item by choosing from one of four answer options from 0 to 3 with higher scores indicating a greater severity of symptom. For scoring, first each subscale score is calculated by finding the mean score of items within the subscale section, subtracting 1, and multiplying that by 100/3. Next, the subscale scores are summed to determine the overall UDI score with possible scores ranging from 0-300. High scores indicate greater symptoms severity.

SECONDARY OUTCOMES:
Incontinence Impact Questionnaire Short Form (IIQ-7) | Change from Baseline IIQ-7 score to 8 weeks and 6 months post-intervention
  Validated short-form version of the Incontinence Impact Questionnaire used to describe incontinence-related quality of life. It consists of 7 items assessing four general areas including travel, social, emotional, and physical activities. For each item, the subject responds by choosing from one of four answer options from 0 to 3 with higher scores indicating a greater severity of symptom. Scores are generated by finding the mean score for each item and multiplying that by 100/3. Higher scores indicate greater negative impact on quality of life.
Urge Urinary Incontinence Episode Frequency on a Three-Day Voiding Diary | Change from Baseline urge urinary incontinence episode frequency to 8 weeks and 6 months post-intervention
  A voiding diary is considered standard of care in the work-up of a patient with incontinence to better characterize real-life drinking and voiding habits. The number of urge urinary incontinence episodes is determined by adding up the incontinence episodes recorded by the patient that were associated with an urge to get to the bathroom. More incontinence episodes means a greater severity of incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Stachowicz, MD, Principal Investigator — Urogynecology Fellow
Locations (1):
- The Christ Hospital, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Milsom I, Coyne KS, Nicholson S, Kvasz M, Chen CI, Wein AJ. Global prevalence and economic burden of urgency urinary incontinence: a systematic review. Eur Urol. 2014 Jan;65(1):79-95. doi: 10.1016/j.eururo.2013.08.031. Epub 2013 Aug 27. PMID 24007713
- [Background] Monteiro S, Riccetto C, Araujo A, Galo L, Brito N, Botelho S. Efficacy of pelvic floor muscle training in women with overactive bladder syndrome: a systematic review. Int Urogynecol J. 2018 Nov;29(11):1565-1573. doi: 10.1007/s00192-018-3602-x. Epub 2018 Apr 11. PMID 29644384
- [Background] Kammerer-Doak D, Rizk DE, Sorinola O, Agur W, Ismail S, Bazi T. Mixed urinary incontinence: international urogynecological association research and development committee opinion. Int Urogynecol J. 2014 Oct;25(10):1303-12. doi: 10.1007/s00192-014-2485-8. Epub 2014 Aug 5. PMID 25091925
- [Background] Lamin E, Parrillo LM, Newman DK, Smith AL. Pelvic Floor Muscle Training: Underutilization in the USA. Curr Urol Rep. 2016 Feb;17(2):10. doi: 10.1007/s11934-015-0572-0. PMID 26757904
- [Background] Rosenblatt P, Pulliam S, McKinney J, Sutherland R, Iglesias R. The leva incontinence system for the treatment of mild to moderate urinary incontinence: A pilot study. Female Pelvic Med Reconstr Surg.
- [Background] Shumaker SA, Wyman JF, Uebersax JS, McClish D, Fantl JA. Health-related quality of life measures for women with urinary incontinence: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program in Women (CPW) Research Group. Qual Life Res. 1994 Oct;3(5):291-306. doi: 10.1007/BF00451721. PMID 7841963
- [Background] Uebersax JS, Wyman JF, Shumaker SA, McClish DK, Fantl JA. Short forms to assess life quality and symptom distress for urinary incontinence in women: the Incontinence Impact Questionnaire and the Urogenital Distress Inventory. Continence Program for Women Research Group. Neurourol Urodyn. 1995;14(2):131-9. doi: 10.1002/nau.1930140206. PMID 7780440
- [Background] Dyer KY, Xu Y, Brubaker L, Nygaard I, Markland A, Rahn D, Chai TC, Stoddard A, Lukacz E; Urinary Incontinence Treatment Network (UITN). Minimum important difference for validated instruments in women with urge incontinence. Neurourol Urodyn. 2011 Sep;30(7):1319-24. doi: 10.1002/nau.21028. Epub 2011 May 11. PMID 21563210
- [Background] Jimenez-Cidre MA, Lopez-Fando L, Esteban-Fuertes M, Prieto-Chaparro L, Llorens-Martinez FJ, Salinas-Casado J, Castro-Diaz D, Muller-Arteaga C, Adot-Zurbano JM, Rodriguez-Escobar F, Gutierrez C, Arlandis-Guzman S, Bonillo-Garcia MA, Madurga-Patuel B, Leva-Vallejo M, Franco de Castro A, Peri-Cusi L, Conejero-Sugranes J, Jimenez-Calvo J, Rebollo P, Mora A. The 3-day bladder diary is a feasible, reliable and valid tool to evaluate the lower urinary tract symptoms in women. Neurourol Urodyn. 2015 Feb;34(2):128-32. doi: 10.1002/nau.22530. Epub 2013 Nov 22. PMID 24264859
- [Background] Hundley AF, Wu JM, Visco AG. A comparison of perineometer to brink score for assessment of pelvic floor muscle strength. Am J Obstet Gynecol. 2005 May;192(5):1583-91. doi: 10.1016/j.ajog.2004.11.015. PMID 15902162
- [Background] Brink CA, Sampselle CM, Wells TJ, Diokno AC, Gillis GL. A digital test for pelvic muscle strength in older women with urinary incontinence. Nurs Res. 1989 Jul-Aug;38(4):196-9. PMID 2748352